CLINICAL TRIAL: NCT06060457
Title: A Phase 3, Randomized, Observer-Blind Study to Evaluate Safety, Tolerability, and Immunogenicity of mRNA-1345, an mRNA Vaccine Targeting Respiratory Syncytial Virus, When Coadministered With a High-Dose, Quadrivalent Seasonal Influenza Vaccine in Adults ≥65 Years of Age
Brief Title: A Study to Evaluate the Safety and Immune Response of mRNA-1345, a Vaccine Targeting Respiratory Syncytial Virus (RSV), When Co-administered With a Fluzone HD, in Adults ≥65 Years of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: mRNA-1345-P304
Record Dates: First submitted 2023-09-23; First posted 2023-09-29 (Actual); Results first posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Respiratory Syncytial Virus
Keywords: Viral Diseases; Messenger RNA; Moderna; mRNA-1345; Respiratory syncytial virus; Vaccines; RSV Vaccine
MeSH Terms: conditions — Virus Diseases | interventions — mRNA-1345 respiratory syncytial virus vaccine; Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fluzone HD + mRNA-1345 (Experimental): Participants will receive Fluzone HD + mRNA-1345 by intramuscular (IM) injection on Day 1 followed by placebo by IM injection on Day 22.
  Interventions: Biological: Placebo; Biological: mRNA-1345; Biological: Fluzone HD
- Fluzone HD Followed by mRNA-1345 (Experimental): Participants will receive Fluzone HD + placebo by IM injection on Day 1 followed by mRNA-1345 by IM injection on Day 22.
  Interventions: Biological: Placebo; Biological: mRNA-1345; Biological: Fluzone HD

INTERVENTIONS:
Biological: Placebo — 0.9% sodium chloride (normal saline) injection
Biological: mRNA-1345 — Suspension for injection
Biological: Fluzone HD — Suspension for injection

SUMMARY:
The main purpose of this study is to evaluate the safety and immunogenicity of mRNA-1345 RSV vaccine when coadministered with a high dose (HD) quadrivalent seasonal influenza vaccine (Fluzone HD) in adults ≥65 years of age. The study will examine the impact of Fluzone HD on the immune response to mRNA-1345 against RSV-A and RSV-B, as well as the impact of mRNA-1345 on the immune response to Fluzone HD against 4 vaccine-matched Influenza A and B strains.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants may have one or more chronic medical diagnoses, but should be medically stable as assessed by:

  * Absence of changes in medical therapy within 60 days of Day 1 due to treatment failure or toxicity,
  * Absence of serious or significant medical events within 30 days of Day 1, and
  * Absence of known, current, and life-limiting diagnoses which, in the opinion of the Investigator, would make completion of the protocol unlikely.
* A participant assigned female at birth is eligible to participate if they are postmenopausal or not a person of childbearing potential.

Key Exclusion Criteria:

* Close contact with someone with laboratory-confirmed influenza and/or RSV infection or with someone who has been treated with antiviral therapies for influenza (for example, Tamiflu®) within the past 5 days prior to Day 1.
* Reported history of congenital or acquired immunodeficiency, immunosuppressive condition or immune-mediated disease, asplenia, or recurrent severe infections.
* Participant has tested positive for influenza or RSV by local health authority-approved testing methods ≤6 months prior to Day 1.
* Participant has received or plans to receive any vaccine authorized or approved by a local health agency ≤28 days prior to study injections (Day 1 and Day 22) or plans to receive a vaccine authorized or approved by a local health agency within 28 days after study injections.
* Participant has received a seasonal influenza vaccine or any other investigational influenza vaccine ≤6 months prior to Day 1.
* Participant has received any RSV vaccine (authorized/approved by local health agency or investigational) prior to Day 1.

Note: Other protocol-defined inclusion and/or exclusion criteria may apply.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 1900 (Actual)
Dates: Start 2023-09-25 (Actual); Primary Completion 2024-06-07 (Actual); Study Completion 2024-06-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (34):
- United States (34):
  - Scottsdale Clinical Trials, Scottsdale, Arizona
  - Headlands Research, Inc., Scottsdale, Arizona
  - West Coast Research LLC, Dublin, California
  - Artemis Institute for Clinical Research, Riverside, California
  - Peninsula Research Associates (PRA), Rolling Hills Estates, California
  - Acclaim Clinical Research, San Diego, California
  - Neoclinical Research, Hialeah, Florida
  - Health Awareness INC, Jupiter, Florida
  - South Florida Research Center, Inc., Miami, Florida
  - Suncoast Research Associates, LLC, Miami, Florida
  - Headlands Research - Orlando, Orlando, Florida
  - New Tampa Health, Inc, Tampa, Florida
  - Clinical Research Atlanta/Headlands, Stockbridge, Georgia
  - Bingham Memorial Hospital, Blackfoot, Idaho
  - DM Clinical Research- River Forest, River Forest, Illinois
  - Velocity Clinical Research-Baton Rouge, Baton Rouge, Louisiana
  - DelRicht Research @ Neighborhood Health, Prairieville, Louisiana
  - DM Clinical Research - Brookline, Brookline, Massachusetts
  - DM Clinical Research - Southfield, Southfield, Michigan
  - Delricht Research at Gulfport Memorial, Gulfport, Mississippi
  - Delricht Research, Springfield, Missouri
  - Be Well Clinical Studies, LLC, Lincoln, Nebraska
  - Velocity Clinical Research-Norfolk, Norfolk, Nebraska
  - Trial Management Associates, LLC, Wilmington, North Carolina
  - Synexus AES - Akron, Akron, Ohio
  - Centricity Research, Columbus, Ohio
  - Delricht Tate, Tulsa, Oklahoma
  - DM Clinical Research - Philadelphia, Philadelphia, Pennsylvania
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - Delricht Moyer, Hendersonville, Tennessee
  - DM Clinical Research - Houston, Houston, Texas
  - DELRICHT RESEARCH at ZOMNIR FAMILY MEDICINE, McKinney, Texas
  - Javara Inc. /Privia Medical Group Gulf Coast, PLLC, Sugar Land, Texas
  - DM Clinical Research, Tomball, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Fluzone HD + mRNA-1345 Followed by Placebo: Participants received Fluzone High Dose (HD) + mRNA-1345 by intramuscular (IM) injection on Day 1 followed by placebo by IM injection on Day 22.
- Fluzone HD + Placebo Followed by mRNA-1345: Participants received Fluzone HD + placebo by IM injection on Day 1 followed by mRNA-1345 by IM injection on Day 22.
Period: Overall Study
Arm/Group | Fluzone HD + mRNA-1345 Followed by Placebo | Fluzone HD + Placebo Followed by mRNA-1345
Started | 950 | 950
Received Day 1 Injection | 946 | 947
Received Day 22 Injection | 919 | 911
Safety Set (All randomized participants who received any study intervention. Participants were included in the treatment arm corresponding to the study drug they actually received.) | 947 | 946 (1 participant received wrong injection (Fluzone HD + mRNA-1345 Followed by Placebo) instead of receiving 'Fluzone HD + Placebo Followed by mRNA-1345'.)
Completed | 914 | 909
Not Completed | 36 | 41
Not completed — Adverse Event | 1 | 1
Not completed — Death | 2 | 2
Not completed — Lost to Follow-up | 17 | 19
Not completed — Physician Decision | 0 | 1
Not completed — Protocol Violation | 1 | 1
Not completed — Serious Adverse Reaction (SAR)/Reactogenicity Event | 1 | 1
Not completed — Withdrawal by Subject | 12 | 15
Not completed — Other Than Specified | 2 | 1

BASELINE CHARACTERISTICS:
Population: The Randomized Set included all participants who were randomized in the study, regardless of the participant's treatment status in the study.
Groups:
- Fluzone HD + mRNA-1345 Followed by Placebo: Participants received Fluzone HD + mRNA-1345 by IM injection on Day 1 followed by placebo by IM injection on Day 22.
- Total: Total of all reporting groups
Arm/Group | Fluzone HD + mRNA-1345 Followed by Placebo | Fluzone HD + Placebo Followed by mRNA-1345 | Total
Number analyzed (Participants) | 950 | 950 | 1900
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.7 (4.80) | 70.7 (4.80) | 70.7 (4.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 548 | 530 | 1078
  Male | 402 | 420 | 822
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 209 | 222 | 431
  Not Hispanic or Latino | 728 | 722 | 1450
  Unknown or Not Reported | 13 | 6 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 7 | 2 | 9
  Asian | 13 | 12 | 25
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 187 | 191 | 378
  White | 735 | 738 | 1473
  More than one race | 7 | 3 | 10
  Unknown or Not Reported | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Local and Systemic Adverse Reactions (ARs) Within 7 Days After Day 1 Injection
Description: Solicited ARs were collected in an electronic diary (eDiary). Local ARs: injection site pain, erythema (redness), swelling/induration (hardness); and axillary (underarm) swelling or tenderness ipsilateral to the side of injection. Systemic ARs: fever, headache, fatigue, myalgia, arthralgia, nausea/vomiting, and chills. Note, not all solicited ARs were considered adverse events (AEs). Investigator reviewed whether the solicited AR was also to be recorded as an AE. A Summary of serious AEs (SAEs) and nonserious AEs ("Other"), regardless of causality, is located in the "Reported Adverse Events" section.
Time Frame: Within 7 days after Day 1 injection
Population: Day 1 Solicited Safety Set included all randomized participants who received any study intervention on Day 1 and contributed any solicited ARs data from the time of study injection on Day 1 through the following 6 days. Participants were included in the treatment arm corresponding to the study drug they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluzone HD + mRNA-1345 Followed by Placebo | Fluzone HD + Placebo Followed by mRNA-1345
Number analyzed (Participants) | 947 | 945
Participants | 689 | 547

2. Primary Outcome: Number of Participants With Solicited Local and Systemic ARs Within 7 Days After Day 22 Injection
Description: Solicited ARs were collected in an eDiary. Local ARs: injection site pain, erythema (redness), swelling/induration (hardness); and axillary (underarm) swelling or tenderness ipsilateral to the side of injection. Systemic ARs: fever, headache, fatigue, myalgia, arthralgia, nausea/vomiting, and chills. Note, not all solicited ARs were considered AEs. Investigator reviewed whether the solicited AR was also to be recorded as an AE. A Summary of SAEs and nonserious AEs ("Other"), regardless of causality, is located in the "Reported Adverse Events" section.
Time Frame: Within 7 days after Day 22 injection
Population: Day 22 Solicited Safety Set included all randomized participants who received any study intervention on Day 22 and contributed any solicited ARs data from the time of study injection on Day 22 through the following 6 days. Participants were included in the treatment arm corresponding to the study drug they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluzone HD + mRNA-1345 Followed by Placebo | Fluzone HD + Placebo Followed by mRNA-1345
Number analyzed (Participants) | 919 | 910
Participants | 251 | 557

3. Primary Outcome: Number of Participants With Unsolicited Adverse Events (AEs) Up to 21 Days After Day 1 Injection
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. Any abnormal laboratory test result (hematology, clinical chemistry, or prothrombin time [PT]/partial thromboplastin time [PTT]) or other safety assessment (for example, electrocardiogram, radiological scan, vital sign measurement), including one that worsened from baseline and was considered clinically significant in the medical and scientific judgment of the Investigator was recorded as an AE. A summary of SAEs and all nonserious AEs ("Other"), regardless of causality, is located in the "Reported Adverse Events" section.
Time Frame: Up to 21 days after Day 1 injection
Population: The Safety Set included all randomized participants who received any study intervention. Participants were included in the treatment arm corresponding to the study drug they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluzone HD + mRNA-1345 Followed by Placebo | Fluzone HD + Placebo Followed by mRNA-1345
Number analyzed (Participants) | 947 | 946
Participants | 72 | 72

4. Primary Outcome: Number of Participants With Unsolicited AEs Up to 21 Days After Day 22 Injection
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. Any abnormal laboratory test result (hematology, clinical chemistry, or PT/PTT) or other safety assessment (for example, electrocardiogram, radiological scan, vital sign measurement), including one that worsened from baseline and was considered clinically significant in the medical and scientific judgment of the Investigator was recorded as an AE. A summary of SAEs and all nonserious AEs ("Other"), regardless of causality, is located in the "Reported Adverse Events" section.
Time Frame: Up to 21 days after Day 22 injection
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Fluzone HD + mRNA-1345 Followed by Placebo | Fluzone HD + Placebo Followed by mRNA-1345
Number analyzed (Participants) | 947 | 946
Participants | 60 | 71

5. Primary Outcome: Number of Participants With Medically Attended Adverse Events (MAAEs), Adverse Events of Special Interest (AESIs), Serious Adverse Events (SAEs), and AEs Leading to Discontinuation
Description: A MAAE is an AE that leads to an unscheduled visit to a healthcare practitioner. An AESI is an AE (serious or nonserious) of scientific and medical concern specific to the Sponsor's product or program, for which ongoing monitoring and immediate notification by the Investigator to the Sponsor are required. An SAE was defined as any AE that resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in disability, was a congenital anomaly/birth defect, or was an important medical event. A summary of SAEs and all nonserious AEs ("Other"), regardless of causality, is located in the "Reported Adverse Events" section.
Time Frame: Day 1 through Day 202
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Fluzone HD + mRNA-1345 Followed by Placebo | Fluzone HD + Placebo Followed by mRNA-1345
Number analyzed (Participants) | 947 | 946
Participants
  MAAEs | 194 | 191
  AESIs | 0 | 1
  SAEs | 23 | 33
  AEs Leading to Discontinuation | 3 | 3

6. Primary Outcome: Geometric Mean Titer (GMT) of Serum Respiratory Syncytial Virus Subtype A (RSV-A) and Respiratory Syncytial Virus Subtype B (RSV-B) Neutralizing Antibodies (nAbs)
Description: Antibody values reported as below lower limit of quantification (LLOQ) were replaced by 0.5*LLOQ. Values greater than the upper limit of quantification (ULOQ) were replaced by the ULOQ. LLOQ was 13 international units (IU)/milliliter (mL) and ULOQ was 259061 IU/mL for RSV-A. LLOQ was 10 IU/mL and ULOQ was 112476 for RSV-B.
Time Frame: Day 22 (for Arm 1) and Day 43 (for Arm 2)
Population: The Per-protocol (PP) Set included all randomized participants who received the assigned study intervention dose according to protocol, complied with immunogenicity blood sampling to have a baseline and at least 1 post-injection assessment, and had no important protocol deviations that impacted the immune response. 'Overall number of participants analyzed' = participants evaluable for this endpoint. 'Number analyzed' = participants evaluable for specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Fluzone HD + mRNA-1345 Followed by Placebo | Fluzone HD + Placebo Followed by mRNA-1345
Number analyzed (Participants) | 897 | 858
IU/mL
  RSV-A | 11800.26 [11063.69 to 12585.87] | 18874.12 [17670.37 to 20159.87]
  RSV-B: number analyzed (Participants) | 896 | 842
  RSV-B | 4197.74 [3949.53 to 4461.54] | 6579.15 [6178.21 to 7006.11]
Statistical Analysis 1: Comparison: Fluzone HD + mRNA-1345 Followed by Placebo vs Fluzone HD + Placebo Followed by mRNA-1345; RSV-A: Arm 1 versus Arm 2; Test type: Other; Geometric Mean Ratio (GMR) = 0.625, 95% CI 2-sided [0.570 to 0.686]
Statistical Analysis 2: Comparison: Fluzone HD + mRNA-1345 Followed by Placebo vs Fluzone HD + Placebo Followed by mRNA-1345; RSV-B: Arm 1 versus Arm 2; Test type: Other; GMR = 0.638, 95% CI 2-sided [0.584 to 0.697]

7. Primary Outcome: GMT of Serum Anti-Hemagglutination (HA) Ab Level, as Measured by Hemagglutination Inhibition (HAI) Assay
Description: Influenza A strains included H1N1 and H3N2 and influenza B strains included Austria and Phuket strains. Antibody values reported as below LLOQ were replaced by 0.5*LLOQ. Values greater than the ULOQ were replaced by the ULOQ. LLOQ was 10 and ULOQ was 2560 for Influenza A. LLOQ was 10 and ULOQ was 640 for Influenza B.
Time Frame: Day 22
Population: The PP Set included all randomized participants who received the assigned study intervention dose according to protocol, complied with immunogenicity blood sampling to have a baseline and at least 1 post-injection assessment, and had no important protocol deviations that impacted the immune response. 'Overall number of participants analyzed' = participants evaluable for this endpoint.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Fluzone HD + mRNA-1345 Followed by Placebo | Fluzone HD + Placebo Followed by mRNA-1345
Number analyzed (Participants) | 894 | 880
titer
  Influenza A H1N1 Antibody | 108.11 [99.76 to 117.15] | 124.15 [114.49 to 134.62]
  Influenza A H3N2 Antibody | 198.53 [183.61 to 214.67] | 228.83 [211.50 to 247.58]
  Influenza B Austria Antibody | 105.32 [98.34 to 112.80] | 118.27 [110.37 to 126.74]
  Influenza B Phuket Antibody | 33.17 [31.28 to 35.17] | 34.97 [32.97 to 37.10]

8. Secondary Outcome: Percentage of Participants With Seroresponse for RSV-A and RSV-B nAbs, as Measured by HAI Assay
Description: Seroresponse at a participant level was defined as a change from below the LLOQ to equal or above 4 * LLOQ, or at least a 4-fold increase if baseline was equal to or above the LLOQ. LLOQ was 13 IU/mL and ULOQ was 259061 IU/mL for RSV-A. LLOQ was 10 IU/mL and ULOQ was 112476 for RSV-B.
Time Frame: Baseline to Day 22 (for Arm 1) or Day 43 (for Arm 2)
Population: The PP Set included all randomized participants who received the assigned study intervention dose according to protocol, complied with immunogenicity blood sampling to have a baseline and at least 1 post-injection assessment, and had no important protocol deviations that impacted the immune response. 'Overall number of participants analyzed' = participants evaluable for this endpoint. 'Number analyzed' = participants evaluable for specified category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fluzone HD + mRNA-1345 Followed by Placebo | Fluzone HD + Placebo Followed by mRNA-1345
Number analyzed (Participants) | 897 | 858
percentage of participants
  RSV-A | 64.7 [61.4 to 67.8] | 78.2 [75.3 to 80.9]
  RSV-B: number analyzed (Participants) | 896 | 842
  RSV-B | 48.7 [45.3 to 52.0] | 61.9 [58.5 to 65.2]

9. Secondary Outcome: Geometric Mean Fold-Rise (GMFR) of Postinjection RSV-A and RSV-B nAbs Antibodies for Influenza, as Measured by HAI Assay
Description: 95% CI for GMFR was calculated based on the t-distribution of the differences in the log-transformed values between analysis timepoint and baseline, then back transformed to the original scale for presentation.
Time Frame: Day 22 (for Arm 1) or Day 43 (for Arm 2)
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Fluzone HD + mRNA-1345 Followed by Placebo | Fluzone HD + Placebo Followed by mRNA-1345
Number analyzed (Participants) | 897 | 858
ratio
  RSV-A | 6.49 [6.03 to 6.99] | 10.00 [9.25 to 10.82]
  RSV-B: number analyzed (Participants) | 896 | 842
  RSV-B | 4.08 [3.81 to 4.36] | 5.92 [5.48 to 6.39]

10. Secondary Outcome: Percentage of Participants With ≥2-fold Increase in RSV-A and RSV-B nAbs
Description: ≥2-fold increase from baseline at participant level was defined as a change from below the LLOQ to equal or above 2 * LLOQ, or at least a 2-fold increase if baseline was equal to or above the LLOQ. LLOQ was 13 IU/mL and ULOQ was 259061 IU/mL for RSV-A. LLOQ was 10 IU/mL and ULOQ was 112476 for RSV-B.
Time Frame: Day 22 (Arm 1) or Day 43 (Arm 2)
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fluzone HD + mRNA-1345 Followed by Placebo | Fluzone HD + Placebo Followed by mRNA-1345
Number analyzed (Participants) | 897 | 858
percentage of participants
  RSV-A | 85.4 [82.9 to 87.6] | 93.2 [91.3 to 94.8]
  RSV-B: number analyzed (Participants) | 896 | 842
  RSV-B | 75.4 [72.5 to 78.2] | 83.5 [80.8 to 85.9]

11. Secondary Outcome: Percentage of Participants With Seroconversion, as Measured by HAI Assay
Description: Influenza A strains included H1N1 and H3N2 and influenza B strains included Austria and Phuket strains. Seroconversion at a participant level was defined as a titer ≥1:40 if baseline is < 1:10 or at least a 4-fold increase from baseline if baseline was ≥1:10. Antibody values reported as below LLOQ were replaced by 0.5*LLOQ. Values greater than the ULOQ were replaced by the ULOQ. LLOQ was 10 and ULOQ was 2560 for Influenza A. LLOQ was 10 and ULOQ was 640 for Influenza B.
Time Frame: Day 22
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fluzone HD + mRNA-1345 Followed by Placebo | Fluzone HD + Placebo Followed by mRNA-1345
Number analyzed (Participants) | 894 | 880
percentage of participants
  Influenza A H1N1 Antibody | 56.0 [52.7 to 59.3] | 59.0 [55.6 to 62.2]
  Influenza A H3N2 Antibody | 60.3 [57.0 to 63.5] | 65.8 [62.6 to 68.9]
  Influenza B Austria Antibody | 55.5 [52.2 to 58.8] | 59.1 [55.8 to 62.4]
  Influenza B Phuket Antibody | 31.7 [28.6 to 34.8] | 32.8 [29.7 to 36.1]

12. Secondary Outcome: GMFR of Serum Ab Level, as Measured by HAI Assay
Description: as for outcome 9
Time Frame: Day 22
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Fluzone HD + mRNA-1345 Followed by Placebo | Fluzone HD + Placebo Followed by mRNA-1345
Number analyzed (Participants) | 894 | 880
ratio
  Influenza A H1N1 Antibody | 5.21 [4.76 to 5.71] | 5.78 [5.25 to 6.36]
  Influenza A H3N2 Antibody | 6.20 [5.64 to 6.82] | 7.16 [6.49 to 7.89]
  Influenza B Austria Antibody | 4.87 [4.48 to 5.30] | 5.64 [5.17 to 6.16]
  Influenza B Phuket Antibody | 2.73 [2.56 to 2.90] | 2.88 [2.70 to 3.07]

13. Other Pre Specified Outcome: Number of Deaths Related to Study Drug
Description: A death that occurred during the study or that came to the attention of the investigator during the study was reported to the Sponsor, whether or not it was considered related to study drug. The investigator assessed causality (that is, whether there is a reasonable possibility that the study drug caused the death). The relationship was characterized using the following classifications: Not related: There was not a reasonable possibility of a relationship to the study drug. The temporal sequence of the death relative to administration of the study drug was not reasonable AND/OR the death was more likely explained by a cause other than the study drug. Related: There was a reasonable possibility of a relationship to the study drug. There was evidence of exposure to the study drug. The temporal sequence of the death relative to the administration of the study drug was reasonable. The death was more likely explained by the study drug than by another cause.
Time Frame: Day 1 through Day 202
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Fluzone HD + mRNA-1345 Followed by Placebo | Fluzone HD + Placebo Followed by mRNA-1345
Number analyzed (Participants) | 947 | 946
Participants
  Deaths | 2 | 2
  Deaths related to study drug | 0 | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality and serious adverse events were collected Day 1 up to Day 202. Other (not including serious) unsolicited adverse events were collected up to 21 days after each study injection (that is, Day 1 up to Day 21 for the first injection and Day 22 up to Day 43 for the second injection).
Description: All-cause mortality based on randomization set. SAEs and other (not including serious) AEs based on safety set (all randomized participants who received any study vaccination). Participants included in treatment arm corresponding to study drug they actually received. Per prespecified analysis, all-cause mortality, SAE, and other (not including serious) AE data were collected by arm assignment of "Fluzone HD + mRNA-1345 Followed by Placebo" or "Fluzone HD + Placebo Followed by mRNA-1345".
Arm/Group | Fluzone HD + mRNA-1345 Followed by Placebo | Fluzone HD + Placebo Followed by mRNA-1345
All-Cause Mortality (participants affected / at risk) | 2/950 | 2/950
Serious Adverse Events (participants affected / at risk) | 23/947 | 33/946
Other Adverse Events (participants affected / at risk) | 0/947 | 0/946
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluzone HD + mRNA-1345 Followed by Placebo (N=947) | Fluzone HD + Placebo Followed by mRNA-1345 (N=946)
Bacterial sepsis (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 3 (3)
Pneumonia aspiration (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia influenzal (Infections and infestations) | 0 (0) | 1 (1)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Septic encephalopathy (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Chronic lymphocytic leukaemia stage 1 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Drug abuse (Psychiatric disorders) | 0 (0) | 1 (1)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1)
Lacunar infarction (Nervous system disorders) | 0 (0) | 1 (1)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Toxic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Acute left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 2 (2)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 2 (2)
Bradycardia (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 2 (2)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Fibrin D dimer increased (Investigations) | 1 (1) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 1 (1)
Central cord syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dislocation of vertebra (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Traumatic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Device dislocation (Product Issues) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-07-11): https://cdn.clinicaltrials.gov/large-docs/57/NCT06060457/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-10): https://cdn.clinicaltrials.gov/large-docs/57/NCT06060457/SAP_001.pdf